CLINICAL TRIAL: NCT05271201
Title: Effect of Exercise Intensity on Knee and Ankle Joints' Torque and Functional Mobility in Children With Down's Syndrome: a Randomized Controlled Trial
Brief Title: Exercise Intensity for Down Syndrome Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taif University (Other)
Responsible Party: Principal Investigator, Hatem Allam, Assitant prof., Taif University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 291
Record Dates: First submitted 2022-02-26; First posted 2022-03-08 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2022-02

CONDITIONS: Down Syndrome
MeSH Terms: conditions — Down Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mild intensity group (Experimental): Received mild intensity treadmill training according to Martti Karvonen's formula.
  Interventions: Other: treadmill exercise (mild)
- moderate intensity group (Experimental): Received moderate intensity treadmill training according to Martti Karvonen's formula.
  Interventions: Other: treadmill exercise (moderate)

INTERVENTIONS:
Other: treadmill exercise (mild) — mild intensity treadmill training.
  Arms: mild intensity group
Other: treadmill exercise (moderate) — moderate-intensity treadmill training
  Arms: moderate intensity group

SUMMARY:
The current study aimed to determine the appropriate exercise intensity for the rehabilitation of children with down syndrome.

DETAILED DESCRIPTION:
Two groups of down syndrome children were recruited. one group received mild-intensity treadmill training while the other received moderate-intensity treadmill training. Eccentric knee extensors and ankle plantar flexors peak torques were assessed before and after the intervention. Also, functional mobility was assessed for both groups before and after the intervention. The within and between-subjects effect was used to analyze the obtained data before and after the intervention. isokinetic dynamometer and the time up and go test were used for evaluation.

ELIGIBILITY:
Inclusion Criteria:

* independent walking
* Intelligence quotient range from 40 to 70
* right dominant foot
* body mass index from 50 to 75

Exclusion Criteria:

* chronic diseases
* congenital anomalies
* involved in any competitive sport
* previous injury to the lower limb

Ages: 8 Years to 12 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 34 (Actual)
Dates: Start 2019-12-10 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2020-03-27 (Actual)

PRIMARY OUTCOMES:
knee extensor peak torque | three months
  eccentric normalized peak torque of the knee extensors of the dominant limb.
ankle plantar fexors peak torque | three months
  eccentric normalized peak torque of the ankle plantar flexors of the dominant limb.
functional mobility | three months
  the assessment of the time up and go test

CONTACTS AND LOCATIONS:
Overall Officials: Hatem H Allam, ass. prof., Principal Investigator — Taif University
Locations (1):
- College of Applied Medical Sciemces, Ta'if, Mecca Region, Saudi Arabia